CLINICAL TRIAL: NCT05971082
Title: Risk Factors for Advanced Fibrosis Among Fatty Liver Disease Patients Identified Through Pharese-screening of Miaging Reports
Brief Title: Risk Factors for Advanced Fibrosis Among FLD Patients
Acronym: FLD_FU_HUS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Tiinamaija Tuomi, Chief Physician, Helsinki University Central Hospital
Other Study IDs: FLD_FU_HUS
Record Dates: First submitted 2023-06-29; First posted 2023-08-02 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: NAFLD; Liver Cirrhosis; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood and urine samples, blood DNA and RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Recall study: Recruited individuals aged 20-60 at index imaging date invited for follow-up with liver elastography and fat prosentage measurement
  Interventions: Other: Follow-up

INTERVENTIONS:
Other: Follow-up — Follow-up study of progression/remission of liver disease

SUMMARY:
The investigators investigate the heterogeneity fatty liver disease (FLD) as well as risk factors associated with progression of the liver diseases or development of cardiovascular complication. The overarching aim is to develop a AI-based prediction model that could be integrated into the electronic medical record system.

To identify large numbers of unselected individuals with FLD, the investigators developed a phrase recognition algorithm, which identifies FLD using radiology reports. Within the data lake of Helsinki University Hospital, they identified a large number of individuals with or without FLD. The investigators will now randomly invite 1000-1500 individuals with FLD to a follow-up study including investigation of metabolism and progression of liver disease (elastography, blood tests) as well as gathering life-style information. Register data on previous diagnoses and medication will be used to evaluate cardiovascular disease.

DETAILED DESCRIPTION:
The investigators investigate the heterogeneity fatty liver disease (FLD) as well as risk factors associated with progression of the liver diseases or development of cardiovascular complication. The overarching aim is to develop a AI-based prediction model that could be integrated into the electronic medical record system.

To identify large numbers of unselected individuals with FLD, the investigators developed a phrase recognition algorithm, which identifies FLD using radiology reports. This allows them to study also individuals who have had abdominal imaging for any reason (usually not for suspected liver disease). Within the data lake of Helsinki University Hospital, the investigators identified 61,271 individuals with FLD and 155,521 without. The investigators have obtained national register data on their diagnosed diseases and medication.

The investigators will now invite a random sample of 1000-1500 individuals with FLD (aged 20-60 years at the time of the previous imaging) to a follow-up study. Progression of liver disease will be studied by elastography, measurement of fat content and a blood sample for fibrosis markes (ELF score). The participants' metabolism will be evaluated with several laboraroty tests and an i.v. glucagon tolerance test and amino acid response. Questionnaires will be used to obtain life-style information.

ELIGIBILITY:
Inclusion Criteria:

* Liver imaging results in the Helsinki University Hospital datalake 2010-2018 and a finding of fatty liver disease (without liver cirrhosis)
* Age 25-70 years(20-60 yrs at the time of the index imaging (2010-2018)
* Biobank consent with the Helsinki Biobank to be contacted for possible studies

Exclusion Criteria:

Liver cirrhosis at index imaging date; pregnancy; active treatment for cancer

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will invite a random sample of 1000-1500 individuals with FLD (aged 20-60 years at the time of the previous imaging) to a follow-up study. See eligibility criteria for details.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression of liver disease | 5-15 years
  Proportion of participants who have developed liver fibrosis or steatosis since the index date (in 2010-2018)
remission of fatty liver disease | 5-15 years
  Proportion of participants with remission of fatty liver (= no detectable liver fat) since the index date (in 2010-2018)

CONTACTS AND LOCATIONS:
Overall Officials: Tiinamaija Tuomi, MD, PhD, Study Director — Chief Physician
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
Data can be requested from the HUS University Hospital